CLINICAL TRIAL: NCT01328431
Title: Treating Low-Income Smokers in the Hospital Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Steven Bernstein, Principal Investigator, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0907005437; R01CA141479 (NIH)
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Tobacco Use Cessation; Smoking Cessation; Smoking; Tobacco Use Disorder
Keywords: Tobacco Use Cessation; Smoking Cessation; Nicotine Replacement Therapy; Brief Intervention
MeSH Terms: conditions — Tobacco Use Cessation; Smoking Cessation; Smoking; Tobacco Use Disorder | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Subjects receive a brochure for the state's Smokers' Quitline only.
- SBIRT+NRT (Experimental): Subjects receive a 6 week course of NRT, a motivational Brief Negotiated Interview, and a facilitated referral to the state's Smokers' Quitline.
  Interventions: Other: Brief Intervention with NRT Initiation

INTERVENTIONS:
Other: Brief Intervention with NRT Initiation — Brief Negotiated Interview is a manual-guided therapy designed for the ED setting. The purpose is to assist subjects to change some aspect of their smoking and to decide to start nicotine replacement therapy while in the ED. It combines techniques from motivational interviewing and stages of change. a 6-week supply of nicotine replacement therapy is given in the form of patches and gum and subjects are encouraged to use both concurrently. Patches come in 21 mg, 14 mg, and 7 mg doses and the dosage is determined based on how many cigarettes per day a subject is smoking. All subjects receive 400 pieces of 2 mg nicotine gum. All subjects complete a referral form for the state's Smokers' Quitline which is then faxed directly to the Quitline's vendor.
  Arms: SBIRT+NRT

SUMMARY:
This study will test the effectiveness of an Emergency Department (ED) initiated tobacco intervention which includes counseling and medication. Our proposed intervention combines a Brief Negotiated Interview (BNI) with initiation of nicotine patch and gum in the ED, as well as a faxed referral to the state's Smokers' Quitline. A 6 week supply of nicotine patches and nicotine gum are provided to subjects in the intervention arm. Subjects randomized to the control arm will receive a brochure from the state's Smokers' Quitline only.

The primary hypothesis is that the intervention will be superior to the control condition in reducing self-reported and biochemically verified 7-day tobacco abstinence at 3 months.

DETAILED DESCRIPTION:
Of the nation's 45 million adult smokers, nearly 20 million visit hospital emergency departments (EDs) each year. ED patients, particularly smokers, are disproportionately low-income, with limited access to traditional primary care settings. Patients presenting to the ED with a tobacco-related trigger event, like an asthma attack, may be experiencing a "teachable moment." Thus, the ED may be an ideal location in which to identify smokers and initiate treatment for tobacco dependence. Initial pilot research by our group has demonstrated the feasibility of ED-based brief interventions for smokers. Based on our feasibility studies, the Institute of Medicine 2006 report on tobacco and the 2008 US Public Health Service guidelines now list EDs as appropriate loci for tobacco control efforts. This study aims to test the efficacy of an ED-initiated tobacco intervention which includes counseling and medication. The intervention-Screening, Brief Intervention, and Referral to Treatment (SBIRT)-uses a form of motivational interviewing known as the Brief Negotiation Interview (BNI). Our proposed intervention combines a BNI with initiation of nicotine replacement therapy (NRT) and a fax referral to the state Smokers' Quitline during the ED visit. A 6-week starter kit of NRT (patch and/or gum, tailored to level of addiction and patient preference) will be provided with written materials. The initial dose of NRT will be given in the ED. A trained nurse will administer the booster intervention via telephone 3 days post-visit. The SBIRT+NRT arm will be compared to standard care (SC), which consists of written materials only, in a controlled trial of 778 smokers age 18 years or older randomized in a 1:1 fashion.

The primary hypothesis is that SBIRT+NRT will be superior to SC in reducing self-reported and biochemically verified 7-day tobacco abstinence at 3 months. Secondary hypotheses include: (1) Patients with a tobacco related diagnosis for the ED visit will have a higher cessation rate than patients without a tobacco related diagnosis, and (2) Patients who believe their ED visit is smoking-related will have a higher quit rate than others. The investigators will conduct a cost benefit analysis of the interventions. Follow-up assessments at 1, 3 and 12 months will combine self-report with in-person carbon monoxide testing at 3 months for smokers who assert abstinence via phone. Expansions of the proposed project as compared to earlier studies include: 1) initiation of NRT during the ED visit; 2) provision of multiple forms of NRT; 3) a proactive referral made to the Quitline; 4)a credible control condition with minimal baseline assessment, to avoid the assessment reactivity seen in similar ED studies; and 5) an economic analysis of the tested interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Speaks English
* Willing and able to give informed consent
* >100 cigarettes lifetime
* Current daily or some day smoker
* Smokes > 5 cigarettes/day
* Medicaid or self-pay insurance

Exclusion Criteria:

* Too ill or unable to consent
* Not interested in study participation
* Not interested in quitting
* Pregnant, nursing, or trying to conceive
* Current use of tobacco cessation products (patch, gum, inhaler, nasal spray, lozenge, e-cigarette)
* Actively psychotic or mentally ill
* Leaving ED against medical advice
* Investigator discretion
* Lives outside of New Haven County
* Does not have phone with CT area code
* In police custody
* History of allergic reaction to nicotine replacement products
* Currently receiving formal tobacco dependence tx
* Currently taking Zyban, Wellbutrin (bupropion) or Chantix(varenicline)
* Resides in an extended care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Bernstein, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Standard Care | SBIRT+NRT
Started | 390 | 390
Completed | 390 | 388 (Two subjects enrolled in study twice. Protocol violation.)
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2
Period: 1 Month (1M)
Arm/Group | Standard Care | SBIRT+NRT
Started | 390 | 388
Completed | 335 | 330
Not Completed | 55 | 58
Not completed — Lost to Follow-up | 55 | 58
Period: 3 Month (3M)
Arm/Group | Standard Care | SBIRT+NRT
Started | 390 (Attempted to contact all subjects for 3M follow-up, regardless of whether they completed 1M.) | 388 (Attempted to contact all subjects for 3M follow-up, regardless of whether they completed 1M.)
Completed | 313 | 316
Not Completed | 77 | 72
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 75 | 70
Period: 12 Month (12M)
Arm/Group | Standard Care | SBIRT+NRT
Started | 388 (Attempted to contact all subjects at 12M follow-up. Deceased subjects excluded.) | 386 (Attempted to contact all subjects at 12M follow-up. Deceased subjects excluded.)
Completed | 304 | 289
Not Completed | 84 | 97
Not completed — Death | 2 | 6
Not completed — Lost to Follow-up | 82 | 91

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | SBIRT+NRT | Total
Number analyzed (Participants) | 390 | 388 | 778
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 6
  Between 18 and 65 years | 384 | 376 | 760
  >=65 years | 2 | 10 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 218 | 407
  Male | 201 | 170 | 371

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Verification of Tobacco Abstinence
Description: Biochemical verification means a breathalyzer reading for carbon monoxide.
Time Frame: 3 months after enrollment
Population: This is the # of participants in each group.
Measure: Number; unit: participants
Arm/Group | Standard Care | SBIRT+NRT
Number analyzed (Participants) | 388 | 386
participants | 19 [1 to 30] | 47 [1 to 33]

2. Primary Outcome: Self-report of Tobacco Abstinence or Reduction
Description: Questionnaires to assess self reported tobacco abstinence
Time Frame: 3 months
Population: This is the # of participants in each group.
Measure: Number; unit: participants
Arm/Group | Standard Care | SBIRT+NRT
Number analyzed (Participants) | 388 | 386
participants | 34 | 63

3. Secondary Outcome: Self-reported Tobacco Reduction or Abstinence
Description: self-report questionnaires are completed over the phone to assess reduction in cigarette use or abstinence from cigarette use.
Time Frame: 1 month post enrollment
Reporting Status: Not Posted

4. Secondary Outcome: Health Care Service Utilization
Description: A version of the Treatment Services Review (TSR) will be used to assess health care utilization during follow-ups. The TSR is a self-report instrument that asks about hospitalizations, emergency room visits, and outpatient medical and psychiatric care. The version used in this study also asks about how often the subject called the CT Smoker's Quitline, use of NRT or other medications for smoking cessation, and participation in other smoking cessation treatments.
Time Frame: 1 month post enrollment
Reporting Status: Not Posted

5. Secondary Outcome: Self-reported Tobacco Reduction or Abstinence
Description: as for outcome 3
Time Frame: 12 months post enrollment
Reporting Status: Not Posted

6. Secondary Outcome: Health Care Service Utilization
Description: as for outcome 4
Time Frame: 3 months post enrollment
Reporting Status: Not Posted

7. Secondary Outcome: Health Care Service Utilization
Description: as for outcome 4
Time Frame: 12 months post enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: No adverse events reported during the course of the study
Arm/Group | Standard Care | SBIRT+NRT
Serious Adverse Events (participants affected / at risk) | 0/390 | 0/388
Other Adverse Events (participants affected / at risk) | 0/390 | 0/388

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No